CLINICAL TRIAL: NCT02369770
Title: Sensory-Motor Rehabilitation Post Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Principal Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00080466
Record Dates: First submitted 2015-02-07; First posted 2015-02-24 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Acute Stroke
Keywords: Acute Stroke; Robotic therapy; Ankle impairment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Subjects in the Study group will receive stretching and active movement training with robotic guidance and intelligent control
  Interventions: Device: stretching and active movement training
- Control group (Experimental): Subjects in the Control group will receive stretching and active movement training without robotic guidance.
  Interventions: Device: stretching and active movement training

INTERVENTIONS:
Device: stretching and active movement training — A portable rehabilitation robot will be used to strongly or gently move the impaired ankle joint back and forth. Then subjects will be asked to use muscles to move the ankle with or without the robotic guidance depending on which group the subjects are in.

SUMMARY:
Early after stroke, patients often have significant motor impairment and sensory deficit. Evidence has demonstrated heightened plasticity and significant recovery in the acute phase (first months) post stroke but there has been a lack of effective and practical protocols and devices for early intensive sensorimotor therapy.This research study will conduct a randomized clinical trial of an intensive motor-sensory rehabilitation on patients with acute stroke using a wearable rehabilitation robot. The primary aims are to facilitate sensorimotor recovery, reduce ankle impairments, and improve balance and gait functions. This clinical trial will be conducted on the Study and Control groups of acute stroke survivors.

DETAILED DESCRIPTION:
The study will investigate an early intensive rehabilitation in acute stroke for motor relearning, reducing ankle impairments and improving balance and mobility/locomotion functions.

The acute stroke survivor will be randomly placed into two groups. Subjects in the Study group will receive robot-aided motor relearning under real-time feedback, stretching under intelligent control, sensory stimulation, and active movement training with interactive games. Subjects in the Control group will receive passive movement in the middle ROM without intelligent stretching and active movement training without robotic guidance.

For both groups, the therapeutic training will be conducted during 5 hourly sessions (including breaks/transitions between tasks) each week over about 3-week hospital stay. Both groups will also receive the standard of care in the hospital and rehabilitation service. Treatment outcome measures will be obtained through blinded assessments and evaluated before and after training involving biomechanical, neuromuscular and clinical outcome measures. Carry-over effects will be further evaluated 1 month after the treatment ends.

Aim 1: To evaluate biomechanical and neuromuscular changes as defined by the passive and active range of motion (ROM), flexor-extensor muscle strength, joint stiffness, proprioception and reflex excitability, and compare these measures between the two groups. The biomechanical and neuromuscular outcome measures will be obtained through blinded assessments and evaluated before and after training using the wearable rehabilitation robot.

Hypothesis 1: Robot-guided motor relearning, stretching and active movement training (Study group) will improve the biomechanical and neuromuscular outcome measures more than those of the Control group.

Aim 2: To evaluate the clinical outcome measures as defined by Fugl-Meyer score (lower extremity), modified Ashworth scale, Berg balance scale, 10 meter walk test, and to compare between the Study and Control groups.

Hypothesis 2: The Study group will improve the clinical outcome measures more than the Control group.

ELIGIBILITY:
Inclusion Criteria:

1. First time unilateral acute stroke, hemorrhagic or ischemic, 24 hours after admission in hospital to 1 year post stroke.
2. Hemiplegia or hemiparesis
3. Age 18-80
4. Ankle impairments

Exclusion Criteria:

1. No impairment or very mild ankle impairment of ankle.
2. Unstable medical conditions that interferes with ability to training and exercise.
3. Severe cardiovascular disorders that interfere with ability to perform moderate movement exercises.
4. Cognitive impairment or aphasia with inability to follow instructions
5. Pressure ulcer, recent surgical incision or active skin disease with open wounds present below knee of treated limb
6. Severe pain in legs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Fugl-Meyer Lower Extremity (FMLE) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The assessment is a measure of lower extremity (LE) motor and sensory impairments.

SECONDARY OUTCOMES:
Changes of active range of motion (AROM) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  AROM will be measured in degrees in the ankle joint while subjects use the muscles to move the ankle.
Changes of passive range of motion (PROM) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  PROM will be measured in degrees in the ankle joint while the robot moves the ankle of the subject strongly.
Changes of ankle strength | At the beginning and end of 3-week training, and 1 month after the treatment ends
  Strength of the ankle flexor-extensor muscle will be measured in Newton
Changes of ankle stiffness | At the beginning and end of 3-week training, and 1 month after the treatment ends
  Spasticity will be measured by the resistance torque in Newton-meter under controlled movement at each joint.
Changes of Modified Ashworth Scale (MAS) | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The Modified Ashworth Scale is the most widely used assessment tool to measure resistance to limb movement in a clinic setting. Scores range from 0-4, with 6 choices. 0 (0) - No increase in muscle tone; 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension; 1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM (range of movement); 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved; 3 (4) - Considerable increase in muscle tone passive, movement difficult; 4 (5) - Affected part(s) rigid in flexion or extension.
Changes of Berg Balance Scale | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The Berg balance scale is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Changes of 10 meter Walk Test | At the beginning and end of 3-week training, and 1 month after the treatment ends
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albert SJ, Kesselring J. Neurorehabilitation of stroke. J Neurol. 2012 May;259(5):817-32. doi: 10.1007/s00415-011-6247-y. Epub 2011 Oct 1. PMID 21964750
- [Background] Bernhardt J, Chan J, Nicola I, Collier JM. Little therapy, little physical activity: rehabilitation within the first 14 days of organized stroke unit care. J Rehabil Med. 2007 Jan;39(1):43-8. doi: 10.2340/16501977-0013. PMID 17225037
- [Background] Bernhardt J, Dewey H, Thrift A, Donnan G. Inactive and alone: physical activity within the first 14 days of acute stroke unit care. Stroke. 2004 Apr;35(4):1005-9. doi: 10.1161/01.STR.0000120727.40792.40. Epub 2004 Feb 26. PMID 14988574
- [Background] Chung SG, van Rey E, Bai Z, Rymer WZ, Roth EJ, Zhang LQ. Separate quantification of reflex and nonreflex components of spastic hypertonia in chronic hemiparesis. Arch Phys Med Rehabil. 2008 Apr;89(4):700-10. doi: 10.1016/j.apmr.2007.09.051. PMID 18374001
- [Background] Chung SG, Van Rey E, Bai Z, Roth EJ, Zhang LQ. Biomechanic changes in passive properties of hemiplegic ankles with spastic hypertonia. Arch Phys Med Rehabil. 2004 Oct;85(10):1638-46. doi: 10.1016/j.apmr.2003.11.041. PMID 15468024
- [Background] Chen K, Wu YN, Ren Y, Liu L, Gaebler-Spira D, Tankard K, Lee J, Song W, Wang M, Zhang LQ. Home-Based Versus Laboratory-Based Robotic Ankle Training for Children With Cerebral Palsy: A Pilot Randomized Comparative Trial. Arch Phys Med Rehabil. 2016 Aug;97(8):1237-43. doi: 10.1016/j.apmr.2016.01.029. Epub 2016 Feb 20. PMID 26903143
- [Background] Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society; Delgado MR, Hirtz D, Aisen M, Ashwal S, Fehlings DL, McLaughlin J, Morrison LA, Shrader MW, Tilton A, Vargus-Adams J. Practice parameter: pharmacologic treatment of spasticity in children and adolescents with cerebral palsy (an evidence-based review): report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2010 Jan 26;74(4):336-43. doi: 10.1212/WNL.0b013e3181cbcd2f. PMID 20101040
- [Background] Gao F, Grant TH, Roth EJ, Zhang LQ. Changes in passive mechanical properties of the gastrocnemius muscle at the muscle fascicle and joint levels in stroke survivors. Arch Phys Med Rehabil. 2009 May;90(5):819-26. doi: 10.1016/j.apmr.2008.11.004. PMID 19406302
- [Background] Gao F, Ren Y, Roth EJ, Harvey R, Zhang LQ. Effects of repeated ankle stretching on calf muscle-tendon and ankle biomechanical properties in stroke survivors. Clin Biomech (Bristol). 2011 Jun;26(5):516-22. doi: 10.1016/j.clinbiomech.2010.12.003. Epub 2011 Jan 6. PMID 21211873
- [Background] Gao F, Zhang LQ. Altered contractile properties of the gastrocnemius muscle poststroke. J Appl Physiol (1985). 2008 Dec;105(6):1802-8. doi: 10.1152/japplphysiol.90930.2008. Epub 2008 Oct 23. PMID 18948443
- [Background] Jenkins WM, Merzenich MM. Reorganization of neocortical representations after brain injury: a neurophysiological model of the bases of recovery from stroke. Prog Brain Res. 1987;71:249-66. doi: 10.1016/s0079-6123(08)61829-4. No abstract available. PMID 3588947
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Jin D, Ren Y, Chen K, Harvey RL, Roth EJ, Prabhakaran S, and Zhang L-Q. Mobility rehabilitation in acute stroke using a wearable ankle robot. Neuroscience, Chicago, 2015
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Management of Stroke Rehabilitation Working Group. VA/DOD Clinical practice guideline for the management of stroke rehabilitation. J Rehabil Res Dev. 2010;47(9):1-43. No abstract available. PMID 21213454
- [Background] Murphy TH, Corbett D. Plasticity during stroke recovery: from synapse to behaviour. Nat Rev Neurosci. 2009 Dec;10(12):861-72. doi: 10.1038/nrn2735. Epub 2009 Nov 4. PMID 19888284
- [Background] Nudo RJ, Milliken GW. Reorganization of movement representations in primary motor cortex following focal ischemic infarcts in adult squirrel monkeys. J Neurophysiol. 1996 May;75(5):2144-9. doi: 10.1152/jn.1996.75.5.2144. PMID 8734610
- [Background] Ren Y, Wu YN, Yang CY, Xu T, Harvey RL, Zhang LQ. Developing a Wearable Ankle Rehabilitation Robotic Device for in-Bed Acute Stroke Rehabilitation. IEEE Trans Neural Syst Rehabil Eng. 2017 Jun;25(6):589-596. doi: 10.1109/TNSRE.2016.2584003. Epub 2016 Jun 22. PMID 27337720
- [Background] Sanger TD, Delgado MR, Gaebler-Spira D, Hallett M, Mink JW; Task Force on Childhood Motor Disorders. Classification and definition of disorders causing hypertonia in childhood. Pediatrics. 2003 Jan;111(1):e89-97. doi: 10.1542/peds.111.1.e89. PMID 12509602
- [Background] Sawada M, Kato K, Kunieda T, Mikuni N, Miyamoto S, Onoe H, Isa T, Nishimura Y. Function of the nucleus accumbens in motor control during recovery after spinal cord injury. Science. 2015 Oct 2;350(6256):98-101. doi: 10.1126/science.aab3825. Epub 2015 Oct 1. PMID 26430122
- [Background] Selles RW, Li X, Lin F, Chung SG, Roth EJ, Zhang LQ. Feedback-controlled and programmed stretching of the ankle plantarflexors and dorsiflexors in stroke: effects of a 4-week intervention program. Arch Phys Med Rehabil. 2005 Dec;86(12):2330-6. doi: 10.1016/j.apmr.2005.07.305. PMID 16344031
- [Background] Sukal-Moulton T, Clancy T, Zhang LQ, Gaebler-Spira D. Clinical application of a robotic ankle training program for cerebral palsy compared to the research laboratory application: does it translate to practice? Arch Phys Med Rehabil. 2014 Aug;95(8):1433-40. doi: 10.1016/j.apmr.2014.04.010. Epub 2014 May 2. PMID 24792141
- [Background] Waldman G, Yang CY, Ren Y, Liu L, Guo X, Harvey RL, Roth EJ, Zhang LQ. Effects of robot-guided passive stretching and active movement training of ankle and mobility impairments in stroke. NeuroRehabilitation. 2013;32(3):625-34. doi: 10.3233/NRE-130885. PMID 23648617
- [Background] Wu YN, Hwang M, Ren Y, Gaebler-Spira D, Zhang LQ. Combined passive stretching and active movement rehabilitation of lower-limb impairments in children with cerebral palsy using a portable robot. Neurorehabil Neural Repair. 2011 May;25(4):378-85. doi: 10.1177/1545968310388666. Epub 2011 Feb 22. PMID 21343525
- [Background] Wu YN, Ren Y, Goldsmith A, Gaebler D, Liu SQ, Zhang LQ. Characterization of spasticity in cerebral palsy: dependence of catch angle on velocity. Dev Med Child Neurol. 2010 Jun;52(6):563-9. doi: 10.1111/j.1469-8749.2009.03602.x. Epub 2010 Jan 28. PMID 20132137
- [Background] Xerri C, Merzenich MM, Peterson BE, Jenkins W. Plasticity of primary somatosensory cortex paralleling sensorimotor skill recovery from stroke in adult monkeys. J Neurophysiol. 1998 Apr;79(4):2119-48. doi: 10.1152/jn.1998.79.4.2119. PMID 9535973
- [Background] Yang CY, Guo X, Ren Y, Kang SH, Zhang LQ. Position-dependent, hyperexcitable patellar reflex dynamics in chronic stroke. Arch Phys Med Rehabil. 2013 Feb;94(2):391-400. doi: 10.1016/j.apmr.2012.09.029. Epub 2012 Oct 11. PMID 23063880
- [Background] Zhang LQ, Chung SG, Ren Y, Liu L, Roth EJ, Rymer WZ. Simultaneous characterizations of reflex and nonreflex dynamic and static changes in spastic hemiparesis. J Neurophysiol. 2013 Jul;110(2):418-30. doi: 10.1152/jn.00573.2012. Epub 2013 May 1. PMID 23636726
- [Background] Zhang LQ, Rymer WZ. Reflex and intrinsic changes induced by fatigue of human elbow extensor muscles. J Neurophysiol. 2001 Sep;86(3):1086-94. doi: 10.1152/jn.2001.86.3.1086. PMID 11535659
- [Background] Zhang LQ, Wang G, Nishida T, Xu D, Sliwa JA, Rymer WZ. Hyperactive tendon reflexes in spastic multiple sclerosis: measures and mechanisms of action. Arch Phys Med Rehabil. 2000 Jul;81(7):901-9. doi: 10.1053/apmr.2000.5582. PMID 10896002
- [Background] Zhao H, Wu YN, Hwang M, Ren Y, Gao F, Gaebler-Spira D, Zhang LQ. Changes of calf muscle-tendon biomechanical properties induced by passive-stretching and active-movement training in children with cerebral palsy. J Appl Physiol (1985). 2011 Aug;111(2):435-42. doi: 10.1152/japplphysiol.01361.2010. Epub 2011 May 19. PMID 21596920